CLINICAL TRIAL: NCT04490681
Title: Validation of ERTugliflozin for Inhibiting Cardiac Fibrosis Using Cardiac MRI and Laboratory Parameters in Korean Heart Failure Patients With Nonischemic Cardiomyopathy(VERTICAL)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2020-0484
Record Dates: First submitted 2020-07-20; First posted 2020-07-29 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure With Nonischemic Cardiomyopathy
MeSH Terms: interventions — ertugliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the nature of randomized study, it will be masked to all participants, care providers, investigators, and outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ertugliflozin (Experimental): Ertugliflozin 5mg
  Interventions: Drug: Ertugliflozin
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ertugliflozin — Fixed dose Ertugliflozin (5mg)
  Arms: Ertugliflozin
Drug: Placebo — Placebo group
  Arms: placebo

SUMMARY:
Based on recent studies demonstrating SGLT2 inhibitors' favorable effects on cardiovascular outcomes especially for heart failure, the investigators hypothesize that sodium-glucose co-transporter-2 (SGLT2) inhibitor, ertugliflozin, is effective on reducing cardiac fibrosis in patients with nonischemic cardiomyopathy so the investigators try to examine this hypothesis in a single-center, double-blind, randomized controlled study using cardiac magnetic resonance (CMR).

This study is a prospective, single-center, randomized, double-blind, two arm parallel group, placebo-controlled clinical trial involving patients with nonischemic cardiomyopathy. Patients meeting inclusion criteria without any exclusion criteria will be randomized 1:1 to ertugliflozin or placebo therapy, and cardiovascular functional assessment and clinical event follow-up will be undertaken.

DETAILED DESCRIPTION:
Subjects : Patients with non-ischemic cardiomyopathy who need medical treatment Procedures : This is a prospective, randomized trial to compare cardiopulmonary motor tests, cardiac MRI including myocardial fibrosis parameters (ECV, etc.), and incidence of various heart failure-related cardiovascular events during the follow-up period between patients with ertugliflozin drug therapy and placebo drug. Patients meeting inclusion criteria without any exclusion criteria will be randomized 1:1 to ertugliflozin (5mg) or placebo therapy. Randomization will be stratified according to presence of diabetes mellitus, and the upper limit of randomized non-DM patients will be set as 36 patients (70%). The estimated enrollment period is 18 months (n=52) and all patients will be followed for 12 months after randomization. Random assignment is performed at random assignment visit (V1) through eCASE web system and following study procedures will be conducted according to the randomization. CMR, Cardiopulmonary exercise test, serum biomarkers, and clinical endpoints will be measured at 3,6,12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must agree to the study protocol and provide written informed consent
* Outpatients ≥ 19 years, <75 years of age, male or female
* Non-diabetic or type 2 DM patients with HbA1c 7.0-10.5%
* Patients with nonischemic cardiomyopathy (LVEF ≤40%)
* Exclusion of ischemic origin cardiomyopathy using coronary angiography or CT angiography or SPECT scan (e.g. significant stenosis of proximal LAD or left main & myocardial infarction)
* Dyspnea of NYHA functional class II or III
* NT-proBNP ≥ 400 pg/ml (≥ 900 pg/ml if atrial fibrillation or atrial flutter)
* Titration of HF medications should be completed and patients must take a stable, optimized dose of a β-blocker and an ACE inhibitor (or ARB or ARNI if indicated) for at least 4 weeks prior to study entry

Exclusion Criteria:

* History of hypersensitivity or allergy to the study drug, drugs of similar chemical classes, or SGLT-2 as well as known or suspected contraindications to the study drug
* Current use or prior use of a SGLT-2 inhibitor or combined SGLT-1 and 2 inhibitor
* Known history of angioedema
* Current acute decompensated heart failure or dyspnea of NYHA functional class IV
* Medical history of hospitalization within 6 weeks
* Acute coronary syndrome, stroke, major CV surgery, PCI within 3 months
* Substantial myocardial ischemia requiring coronary revascularization therapy or a plan of coronary revascularization within 6 months
* A plan of heart transplantation or implantation of cardiac resynchronization therapy
* Symptomatic hypotension and/or a SBP < 95 mmHg at screening
* Estimated GFR < 30 mL/min/1.73m2
* History of ketoacidosis
* Symptomatic peripheral artery disease and history of lower limb amputation
* Evidence of hepatic disease as determined by any one of the following: AST or ALT values exceeding 3 x upper limit of normal (ULN) at screening visit (Visit 0), history of hepatic encephalopathy, history of esophageal varices, or history of portacaval shunt.
* History of severe pulmonary disease
* Significant mitral & aortic valve disease (e.g. moderate to severe, severe degree)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using a barrier method plus a hormonal method
* Pregnant or nursing (lactating) women
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the investigator, would preclude safe completion of the study

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The ECV value change in CMR after Drug (Ertugliflozin or Placebo) administration | Baseline
  The ECV value change in MRI from baseline to End of trial (48 weeks)
The ECV value change in CMR after Drug (Ertugliflozin or Placebo) administration | 48 Weeks after drug administration
  The ECV value change in MRI from baseline to End of trial (48 weeks)

SECONDARY OUTCOMES:
CMR parameters : ECV (%) | baseline
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : ECV (%) | 12 weeks after drug administration
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : ECV (%) | 48 weeks after drug administration
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : Native T1 (ms) | baseline
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : Native T1 (ms) | 12 weeks after drug administration
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : Native T1 (ms) | 48 weeks after drug administration
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : left & right ventricular (LV & RV) mass index (g/m2) | Baseline
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : left & right ventricular (LV & RV) mass index (g/m2) | 12 weeks after drug administration
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : left & right ventricular (LV & RV) mass index (g/m2) | 48 weeks after drug administration
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : LV & RV ejection fraction (%) | Baseline
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : LV & RV ejection fraction (%) | 12 weeks after drug administration
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : LV & RV ejection fraction (%) | 48 weeks after drug administration
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : LV & RV end-systolic volume, LV & RV end-diastolic volume (ml) | Baseline
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : LV & RV end-systolic volume, LV & RV end-diastolic volume (ml) | 12 weeks after drug administration
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : LV & RV end-systolic volume, LV & RV end-diastolic volume (ml) | 48 weeks after drug administration
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : cine-base cardiac strain (%) | Baseline
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : cine-base cardiac strain (%) | 12 weeks after drug administration
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
CMR parameters : cine-base cardiac strain (%) | 48 weeks after drug administration
  CMR parameters : the changes of myocardial fibrosis markers (ECV, Native T1), ventricular muscle mass marker (left & right ventricular (LV & RV) mass index), ventricular functional markers (LV & RV ejection fraction, cine-base cardiac strain), and ventricular remodeling markers (LV & RV end-systolic volume, LV & RV end-diastolic volume). These parameters represent myocardial fibrotic change, ventricular remodelling, systolic function.
Biomarkers : NT-proBNP, hsTn, soluble ST2, galectin-3, IGFBP7 | baseline
  The change in degree of NT-proBNP, hsTn, soluble ST2, galectin-3, IGFBP7 after drug administration.
Biomarkers : NT-proBNP, hsTn, soluble ST2, galectin-3, IGFBP7 | 12 weeks after drug administration
  The change in degree of NT-proBNP, hsTn, soluble ST2, galectin-3, IGFBP7 after drug administration.
Biomarkers : NT-proBNP, hsTn, soluble ST2, galectin-3, IGFBP7 | 24 weeks after drug administration
  The change in degree of NT-proBNP, hsTn, soluble ST2, galectin-3, IGFBP7 after drug administration.
Biomarkers : NT-proBNP, hsTn, soluble ST2, galectin-3, IGFBP7 | 48 weeks after drug administration
  The change in degree of NT-proBNP, hsTn, soluble ST2, galectin-3, IGFBP7 after drug administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospiatal, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No